CLINICAL TRIAL: NCT02151786
Title: Takepron Intravenous 30 mg Specified Drug-use Survey [Hemostatic Effect/Rebleeding Rate]
Brief Title: Lansoprazole Intravenous 30 mg Specified Drug-use Survey [Hemostatic Effect/Rebleeding Rate]
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 254-011; JapicCTI-142549 (Registry Identifier: JapicCTI); JapicCTI-R160829 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-01

CONDITIONS: Gastric Ulcer, Duodenal Ulcer, Acute Stress Gastritis, and Acute Gastric Mucosal Lesions
Keywords: Pharmacological therapy
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — Lansoprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thirty milligrams of lansoprazole: Thirty milligrams of lansoprazole is mixed in physiological saline (JP) or 5 percent (%) glucose solution for injection (JP) and administered twice daily by drip infusion or dissolved in 20 milliliter (mL) of physiological saline (JP) or 5% glucose solution for injection (JP) and administered twice daily by direct slow intravenous injection.
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole intravenous 30 mg
  Other Names: Takepron Intravenous 30 mg

SUMMARY:
The purpose of this survey is to evaluate the safety (i.e., frequency of adverse events) and efficacy (i.e., hemostatic effect, rate of rebleeding after confirmation of hemostasis) of administration of lansoprazole intravenous 30 milligram (mg) (Takepron Intravenous 30 mg) to a large number of patients in daily medical practice.

DETAILED DESCRIPTION:
This survey was designed to evaluate the safety (i.e., frequency of adverse events) and efficacy (i.e., hemostatic effect, rate of rebleeding after confirmation of hemostasis) of administration of lansoprazole intravenous 30 mg (Takepron Intravenous 30 mg) to a large number of participants in daily medical practice.

For adults, 30 mg of lansoprazole is typically mixed in physiological saline (JP) or 5% glucose solution for injection (JP) and administered twice daily by drip infusion or dissolved in 20 mL of physiological saline (JP) or 5% glucose solution for injection (JP) and administered twice daily by direct slow intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following diseases for whom oral administration is not feasible:

Gastric ulcer, duodenal ulcer, acute stress gastritis, and acute gastric mucosal lesion (all of which should be accompanied by bleeding).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gastric ulcer, duodenal ulcer, acute stress gastritis, and acute gastric mucosal lesions
Sampling Method: Non-Probability Sample
Enrollment: 1120 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 173 investigative site in Japan from 29 January 2007 to 31 March 2010.
Pre-assignment Details: In this study, participants were observed with a historical diagnosis of gastric ulcer or duodenal ulcer or acute stress ulcer or acute gastric mucosal lesion accompanied with bleeding, for whom oral administration of drug was not feasible and were enrolled in single treatment group: Lansoprazole.
Groups:
- Lansoprazole: Lansoprazole 30 milligram (mg), injection or drip infusion, intravenous, twice daily for up to 9 weeks.
Period: Overall Study
Arm/Group | Lansoprazole
Started | 1120
Completed | 1084
Not Completed | 36
Not completed — Unavailability of Case Report Form | 26
Not completed — Outside the Contract Period | 1
Not completed — Randomized, not Treated | 1
Not completed — Unavailability of Information | 8

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Lansoprazole
Number analyzed (Participants) | 1084
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (14.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 350
  Male | 734
Pregnancy Status [Number; unit: participants] — This baseline characteristic was analysed only in female participants.
  participants
    Not Pregnant | 349
    Pregnant | 0
    Unknown | 1
Target Diseases [Number; unit: participants] — Number of participants suffering from different types of ulcer in the study were described in this baseline measure.
  participants
    Gastric Ulcer | 768
    Duodenal Ulcer | 221
    Gastroduodenal Ulcer | 23
    Acute Stress-Induced Ulcer | 8
    Acute Gastric Mucosal Lesion | 60
    Not Provided | 4
Categories of Healthcare [Number; unit: participants] — Participants were categorized as outpatient and inpatient.
  participants
    Outpatient | 11
    Inpatient | 1073
Predisposition to Hypersensitivity [Number; unit: participants] — Participants having tendency to suffer from hypersensitivity were classified in this baseline measure.
  participants
    No | 1042
    Yes | 39
    Unknown | 3
Helicobacter pylori Infection [Number; unit: participants] — Participants diagnosed as positive or negative Helicobacter pylori infection were described in this baseline measure.
  participants
    Negative | 199
    Positive | 434
    Unknown | 451
Alcohol Consumption [Number; unit: participants]
  Alcohol Consumer | 382
  Alcohol Non-Consumer | 547
  Unknown | 155
Smoking Status [Number; unit: participants]
  Smoker | 317
  Non-Smoker | 599
  Unknown | 168
Medical History [Number; unit: participants]
  Have Medical History | 574
  Did not Have Medical History | 510
Breakdown of Medical History [Number; unit: participants] — Participants having more than 1 disease were reported in multiple categories.
  participants
    Peptic Ulcer | 241
    Upper gastrointestinal bleeding | 97
    Cerebrovascular accident | 64
    Malignant Tumor | 59
    Hypertension | 55
    Cardiac Disorders | 55
    Hepatic Dysfunction | 42
    Diabetes Mellitus | 37
    Renal Dysfunction | 13
    Other | 187
Complications [Number; unit: participants]
  Had Complications | 632
  Had no Complications | 452
Breakdown of Complications [Number; unit: participants]
  Hypertension | 206
  Cardiac Disorders | 121
  Diabetes Mellitus | 118
  Hepatic Dysfunction | 115
  Anemia | 78
  Malignant Tumor | 68
  Cerebrovascular Accident | 66
  Renal Dysfunction | 61
  Other | 351
Emotional Stress [Number; unit: participants]
  Had Stress | 129
  Had no Stress | 955
Prior Consumption of Drugs Affecting Coagulation System [Number; unit: participants] — The participants with history of consumption of drugs affecting the coagulation system 1 month prior to study treatment were reported in this baseline measure.
  participants
    No | 758
    Yes | 325
    Unknown | 1
Breakdown of Drugs [Number; unit: participants] — The participants with history of consumption of drugs affecting the coagulation system were categorized in this baseline measure on the basis of drugs which they have taken.
  participants
    Non Steroidal Anti-Inflammatory Drugs | 158
    Platelet aggregation inhibitors | 152
    Anticoagulants | 49
    Steroids | 31
    Other | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to Week 9
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 1084
participants | 35

2. Primary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reactions
Description: Serious adverse drug reactions are defined as serious adverse events (SAEs) which are in the investigator's opinion of causal relationship to the study treatment. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Week 9
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 1084
participants | 9

3. Secondary Outcome: Percentage of Participants With Observed Hemostatic Effect
Description: Hemostatic effect was categorized on the basis of degree of improvement as: markedly improved, moderately improved, slightly improved and poor in the participants with observed hemostatic effect. Efficacy rate was reported as percentage of participants showing efficacy and was calculated as the sum of percentage of number of participants reporting markedly improved + moderately improved + slightly improved divided by the percentage of total number of participants with observed hemostatic effect.
Time Frame: Baseline up to Week 9
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 1052
percentage of participants | 90.3

4. Secondary Outcome: Percentage of Participants With Confirmed Hemostatic Effect
Description: Hemostatic effect was categorized on the basis of degree of improvement as: markedly improved, moderately improved, slightly improved and poor in the participants with confirmed hemostatic effect by endoscopy. Efficacy rate was reported as percentage of participants showing efficacy and was calculated as the sum of percentage of number of participants reporting markedly improved + moderately improved + slightly improved divided by the percentage of total number of participants with confirmed hemostatic effect.
Time Frame: Baseline up to Week 9
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 898
percentage of participants | 91.6

5. Secondary Outcome: Percentage of Participants Who Experienced Rebleeding After Observed Hemostatic Effect
Description: Rebleeding rate was reported as percentage of participants who experienced rebleeding after observed hemostasis and was calculated during the period starting from baseline until the completion of treatment with lansoprazole. It was calculated by dividing the percentage of the number of participants who experienced rebleeding after hemostasis divided by the total number of participants with observed hemostasis.
Time Frame: Baseline up to Week 9
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 819
percentage of participants | 1.1

6. Secondary Outcome: Percentage of Participants Who Experienced Rebleeding After Confirmed Hemostatic Effect
Description: Rebleeding rate was reported as percentage of participants who experienced rebleeding after confirmed hemostasis by endoscopy and was calculated during the period starting from baseline until the completion of treatment with lansoprazole. It was calculated by dividing the percentage of the number of participants who experienced rebleeding after hemostasis divided by the total number of participants with confirmed hemostasis.
Time Frame: Baseline up to Week 9
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 745
percentage of participants | 1.2

7. Secondary Outcome: Percentage of Participants With Observed Hemostatic Effect Who Experienced Rebleeding After the Completion of Treatment
Description: Rebleeding rate was reported as percentage of participants who experienced rebleeding after observed hemostasis and was calculated at 8 weeks after the completion of treatment with lansoprazole. It was calculated by dividing the percentage of the number of participants who experienced rebleeding after hemostasis divided by the total number of participants with observed hemostasis.
Time Frame: Week 8 after the last dose of study drug (Week 17)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 497
percentage of participants | 5.8

8. Secondary Outcome: Percentage of Participants With Confirmed Hemostatic Effect Who Experienced Rebleeding After the Completion of Treatment
Description: Rebleeding rate was reported as percentage of participants who experienced rebleeding after confirmed hemostasis by endoscopy and was calculated at 8 weeks after the completion of treatment with lansoprazole. It was calculated by dividing the percentage of the number of participants who experienced rebleeding after hemostasis divided by the total number of participants with confirmed hemostasis.
Time Frame: Week 8 after the last dose of study drug (Week 17)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 389
percentage of participants | 7.1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 17
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions were collected in this study.
Arm/Group | Lansoprazole
Serious Adverse Events (participants affected / at risk) | 9/1084
Other Adverse Events (participants affected / at risk) | 35/1084
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole (N=1084)
Insomnia (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Depressive Symptom (Psychiatric disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric Haemorrhage (Gastrointestinal disorders) | 4
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
White blood cell count decreased (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lansoprazole (N=1084)
Urinary tract infection (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 1
Depressive symptom (Psychiatric disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Hypogeusia (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 7
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 3
Liver disorder (Hepatobiliary disorders) | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pyrexia (General disorders) | 3
Eosinophil count increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 3
Blood creatinine increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.